CLINICAL TRIAL: NCT02904174
Title: Healthy Living Programme (HLP): Diet, Drug and Fall Prevention for Community-dwelling Frail Older Adults
Brief Title: Healthy Living Programme for Older Adults
Acronym: HLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Pentecostal Church of Hong Kong (Unknown)
Responsible Party: Principal Investigator, TSE Mun Yee Mimi, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-ZJJY
Record Dates: First submitted 2016-09-08; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Frail Older Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Living Programme (Experimental): 6 weeks program, with 45 minutes weekly session over 6 weeks.Week 1 & 2 focused on healthy eating habits including food pyramid, balanced diet for the elderly, food labels, healthy snacks and healthy eating out. Week 3 & 4 were about fall prevention, which included risk factors and complications of fall among older adults, preventive measures, strengthening exercises and aerobic dance. Week 5 & 6 focused on drug management, such as knowledge on commonly used drugs, drug storage, use of analgesics and non-pharmacological pain relief strategies.
  Interventions: Behavioral: Healthy Living Programme

INTERVENTIONS:
Behavioral: Healthy Living Programme — A 6-week Healthy Living Program (HLP) was developed and implemented for all the participants. There was one 45 minutes weekly session over 6 week. Week 1 & 2 focused on healthy eating habits including food pyramid, balanced diet for the elderly, food labels, healthy snacks and healthy eating out. Week 3 & 4 were about fall prevention, which included risk factors and complications of fall among older adults, preventive measures, strengthening exercises and aerobic dance. Week 5 & 6 focused on drug management, such as knowledge on commonly used drugs, drug storage, use of analgesics and non-pharmacological pain relief strategies. Interactive activities such as games, puzzles and question & answer session were included in the group education.

SUMMARY:
Malnutrition, risk of falls and medication incidents are commonly faced by the older adults. This study aimed to provide health education to community-dwelling older adults and to assess the effectiveness of a Healthy Living Program (HLP) to older adults in terms of fall prevention, drug management and healthy eating habits.

DETAILED DESCRIPTION:
This was a single group pre-post trial. Participants aged 60 or above were recruited from the community elderly centres. A 6-week HLP, which included one 45 minutes weekly session, was offered to the participants.

122 participants were recruited. This study shows that the 6-week HLP has a potential to improve the physical well-being of the participants, and to increase their knowledge in diet, drug management and fall prevention.

ELIGIBILITY:
Inclusion Criteria:

* able to communicate and understand Cantonese
* > 1 in frailty score
* members of the Pentecostal Church of Hong Kong

Exclusion Criteria:

* nil

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in subjective happiness level | Baseline, Week 6
  Measured by Subjective Happiness Scale (SHS), which consisted of 4 statements answered on a 7-point Likert scale. Scores for each statement range from 1 to 7 and the scores from the four statements were added, thus the possible range of scores on the SHS is 4 to 28. Higher scores reflect higher levels of subjective happiness.

SECONDARY OUTCOMES:
Change in frailty status | Baseline, Week 6
  Measured by the FRAIL scale, which includes five items: fatigue, resistance, ambulation, illness, and loss of weight. The FRAIL scale ranges from 0-5, with a score of 0 regards as normal, 1-2 as pre-frail and 3-5 as frail.
Change in pain intensity | Baseline, Week 6
  Measured using the numerical rating scale, to assess the presence and intensity of pain among participants, which was presented with 0 referring to no pain and 10 referring to the worst pain imaginable
Change in Generalized pain self-efficacy beliefs | Baseline, Week 6
  Measured by the Pain Self-Efficacy Questionnaire. It consists of 10 statements, and participants were asked to rate their confidence in performing 10 activities or tasks despite experiencing pain, on a 7-point scale.
Change in functional mobility | Baseline, Week 6
  Measured by Timed Up and Go Test. The participants were required to walk a distance of three meters, turn, walk back to the chair and sit down.
Change in hand grip strength | Baseline, Week 6
  Measured using a dynamometer. Participants were seated with arms by the trunk, the elbow flexed to 90 and in a neutral position, and the wrist in slight extension. Participants were told to squeeze the dynamometer as hard as they could
Change in knowledge in healthy eating habits | Baseline, Week 6
  Measured by self-developed questionnaire. Range of score is 0-12, with higher score indicates having more knowledge.
Change in knowledge in drug management | Baseline, Week 6
  Measured by self-developed questionnaire. Range of score is 0-10, with higher score indicates having more knowledge.
Change in knowledge in fall prevention | Baseline, Week 6
  Measured by self-developed questionnaire. Range of score is 0-5, with higher score indicates having more knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Mimi Mun Yee Tse, PhD, Principal Investigator — The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: No